CLINICAL TRIAL: NCT00395928
Title: Chronic and Acute Effect of Smoking on the Left and Right Ventricular Systolic and Diastolic Function in Young Healthy Smokers
Brief Title: Chronic and Acute Effects of Smoking on the Left and Right Ventricular Relaxation in Young Healthy Smokers
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Other Study IDs: KB/126/2001
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2006-11-06 (Estimated); Status verified 2006-11

CONDITIONS: Cardiovascular Diseases
Keywords: heart; echocardiography; diastolic function; left ventricle; right ventricle; cigarette smoking; Smoking; Heart Ventricles; Diastole; Doppler Echocardiography
MeSH Terms: conditions — Cardiovascular Diseases; Cigarette Smoking; Smoking; Heart Murmurs

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Impairment of relaxation, the early phase of ventricular diastole is the first stage of heart diastolic dysfunction. Left ventricular diastolic function can be determined noninvasively by Echo- Doppler - derived mitral valve flow velocities. The addition of pulmonary venous flow pattern enables more accurate assessment of left ventricle diastolic function. The role of the right ventricle in haemodynamic function of the heart is now emphasized. The right ventricle diastolic function can be assess by recording the Doppler tricuspid valve flow pattern. Impaired LV diastolic function usually precedes systolic dysfunction and may cause clinical signs of congestive heart failure. Cigarette smoking is one of the major risk factors for cardiovascular diseases. The aim of the study was to assess left and right ventricular diastolic function in healthy, young and slim smokers before and after smoking one cigarette.

Echocardiographic examination: before and after smoking one cigarette Echocardiographic evaluation of mitral valve flow, pulmonary venous flow, tricuspid valve flow and hepatic vein flow to assess diastolic function of ventricles.

DETAILED DESCRIPTION:
Echocardiographic examination: in left lateral position after 10 minutes rest. The first examination: after a 2-hour non-smoking period, the second: immediately after smoking one cigarette containing 0.9 mg of nicotine. The duration of the second examination: no more than 15 minutes.

Echocardiography equipment: Hewlett-Packard SONOS 2000 (Andover, Massachusetts) imaging system. The transducer's frequency: 2 MHz.

From the apical four chamber view the visualisation of transmitral flow, pulmonary venous flow and transtricuspid flow. From subcostal view the visualisation of right superior hepatic vein and the hepatic vein flow.

ELIGIBILITY:
Inclusion Criteria:

* Smokers smoking over 10 cigarettes per day over the last 5 years
* Body mass index < 25 kg/m2
* Normal blood pressure and normal parameters of echocardiographic examination (wall thickness, left- and right- chamber size, valvular function and left and right ventricular systolic function)
* Normal results of routine physical examination, chest x-ray, standard rest electrocardiogram and routine laboratory tests.

Exclusion Criteria:

* Body mass index > 25 kg/m2
* Abnormal blood pressure
* Abnormal parameters of echocardiographic examination (wall thickness, left- and right- chamber size, valvular function and left and right ventricular systolic function)
* Abnormal results of routine physical examination, chest x-ray, standard rest electrocardiogram and routine laboratory tests.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33
Dates: Start 2001-11; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Danuta Liszewska-Pfejfer, Prof., Study Chair — Internal Medicine and Cardiology Dpt, Warsaw Medical University
Locations (1):
- Internal Medicine and Cardiology Dpt,Institute of Dentistry,Warsaw Medical University, Warsaw, Lindleya 4, Poland

REFERENCES:
- [Background] Oh JK, Appleton CP, Hatle LK, Nishimura RA, Seward JB, Tajik AJ. The noninvasive assessment of left ventricular diastolic function with two-dimensional and Doppler echocardiography. J Am Soc Echocardiogr. 1997 Apr;10(3):246-70. doi: 10.1016/s0894-7317(97)70062-2. PMID 9109691
- [Background] Klein AL, Tajik AJ. Doppler assessment of pulmonary venous flow in healthy subjects and in patients with heart disease. J Am Soc Echocardiogr. 1991 Jul-Aug;4(4):379-92. doi: 10.1016/s0894-7317(14)80448-3. PMID 1910836
- [Background] Voutilainen S, Kupari M, Hippelainen M, Karppinen K, Ventila M, Heikkila J. Factors influencing Doppler indexes of left ventricular filling in healthy persons. Am J Cardiol. 1991 Sep 1;68(6):653-9. doi: 10.1016/0002-9149(91)90360-w. PMID 1877483
- [Background] Alam M, Samad BA, Wardell J, Andersson E, Hoglund C, Nordlander R. Acute effects of smoking on diastolic function in healthy participants: studies by conventional doppler echocardiography and doppler tissue imaging. J Am Soc Echocardiogr. 2002 Oct;15(10 Pt 2):1232-7. doi: 10.1067/mje.2002.124006. PMID 12411910